CLINICAL TRIAL: NCT02271178
Title: Multi-cap for Increase Adherence After Acute Myocardial Infarction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped after interim analysis due to futility.
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Carlos Tajer, MD, Hospital El Cruce
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2014-10-03; First posted 2014-10-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined capsule (Experimental): Combined capsule containing ramipril (5 to 10 mg), atenolol (50 to 100 mg), 100 mg aspirin, 40 mg simvastatin. In follow-up visits doses of atenolol and ramipril capsules may be adjusted according to blood pressure and heart rate.
  Interventions: Other: Combined capsule
- Conventional treatment (Other): Usual therapy
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Combined capsule — Combined capsule containing ramipril (5 to 10 mg), atenolol (50 to 100 mg), 100 mg aspirin, 40 mg simvastatin. In follow-up visits doses of atenolol and ramipril capsules may be adjusted according to blood pressure and heart rate.
  Other Names: Multi-cap.
  Arms: Combined capsule
Other: Conventional therapy — Usual therapy
  Arms: Conventional treatment

SUMMARY:
Patients who survive an acute coronary syndrome are at high risk of recurrent events and death in the first months of evolution. Aspirin, angiotensin-converting enzyme, beta-blockers and statins decrease the risk of recurrent events and death, so are the recommended treatment for most patients who had a heart attack, and adherence to these recommendations is associated better clinical outcome. However, numerous studies show high dropout rate of medical treatment. The cause of nonadherence, common problem in chronic diseases, is multifactorial (economic, cultural, adverse effects), the complexity of the treatment being prescribed a relevant factor as a cause of non-compliance. The investigators goal is to assess whether the simplification of treatment for secondary prevention in a once-daily capsule containing four drugs increased adherence to it, compared to the standard treatment of each drug separately.

The investigators design a controlled, randomized, open, parallel-group clinical study. Patients will be randomized to one of the following treatment regimens:

* Combined-Capsule: capsule containing an adjusted patient combination scheme for secondary prevention of once daily.
* Usual-treatment: each component of the dish separately as is the usual practice.

The primary endpoint is the adherence of the treatment regimen to secondary prevention. For the study was considered adherent to a patient taking at least 80% of medication that belongs in the period.

DETAILED DESCRIPTION:
Sample Size Is estimated according to previous studies adherence to medical treatment 40%, and the objective of the study is to demonstrate an increase in adherence of 25% in absolute terms (40 to 65%) by simplifying the treatment regimen. With a parallel design, a type I error of 5%, a sample of 200 patients would give the study a power of 80% to detect this difference.

A study of this size would also give us increased 80% power to detect a difference of 14 mg / dl in serum cholesterol (estimated standard deviation 30 mg / dl) with an alpha error rate of 5%; and 80% power to detect a difference of 4 mmHg in systolic blood pressure (standard deviation 10 mmHg), also with a type I error of 5%

Procedures

After signing the written informed consent patients will be randomized in a 1:1 ratio, one of the study groups:

* Group 1: Conventional treatment: is a daily tablet of ramipril (5-10 mg / day), atenolol (50-100 mg / day), aspirin 100 mg / day and simvastatin 40 mg / day. The doses of drugs may be increased according to blood pressure and heart rate of patients in follow-up visits.
* Group 2: one capsule containing ramipril (5 to 10 mg), atenolol (50 to 100 mg), 100 mg aspirin, 40 mg simvastatin. In follow-up visits doses of atenolol and ramipril capsules may be adjusted according to blood pressure and heart rate.

All other medications that the patient receives will be determined and adjusted doses as determined by the treating physician.

In patients receiving 100 mg / day and atenolol 10 mg / day of ramipril and require additional treatment to control blood pressure will recommend using thiazide diuretics, calcium channel blockers and alpha-methyldopa, in that order.

All other medications that the patient receives will be determined and adjusted doses as determined by the treating physician.

In patients receiving 100 mg / day and atenolol 10 mg / day of ramipril and require additional treatment to control blood pressure will recommend using thiazide diuretics, calcium channel blockers and alpha-methyldopa, in that order.

The first supply of study medication will be held on discharge from hospital. Patients will be referred for follow-up at 7 days (with an additional 7 days), a month, 3 months and six months (final visit). For visits 2, 3 and 4 be tolerated fifteen (15) days before considering that the patient did not attend the visit.

Randomization After signing the informed consent, patients will be randomized in a 1:1 ratio to receive study treatments.

Randomization was carried out with lists of random numbers generated by computer with a block diagram of 4 and 6. Was also a scheme will use stratified by gender and diabetes.

The mapping is done using consecutive sealed opaque envelopes. To minimize the risk of predicting the next treatment, the envelopes will be handled by the pharmacy staff.

After signing the informed consent was informed pharmacy staff concerned in the study, who will open the appropriate envelope and will be responsible for the preparation and supply of medication (Appendix 1).

Data Anthropometric data, risk factors, cardiovascular history, blood pressure measurements and basal heart rate were collected. All patients will have lab tests including blood count with platelet count, fasting blood glucose, creatinine, urea, electrolytes, liver function tests, total cholesterol, cholesterol bound to high density lipoprotein (HDL) and low density (LDL) , and triglycerides.

Blood pressure and pulse It is measured on the left arm with the subject seated, after 5 minutes of rest. Three blood pressure measurements separated by a minute averaged realized and the last two (discarding the first value). Diastolic blood pressure will be recorded in the fifth Korotkoff sound. Heart rate will be measured by averaging two measurements of 30 seconds; rhythm in patients with atrial fibrillation, two periods of 1 minute averaged. These measurements were repeated at each follow-up visit.

Electrocardiogram ECG were performed at baseline and follow-up, with the subject in supine position after 5 minutes of rest. All are made with automatic ECG 12-lead equipment and will be printed to be analyzed manually.

Laboratory The baseline analysis was performed on admission to the coronary care unit (routine practice), in this analysis is considered basal level of lipids (total cholesterol and fractions) on admission to hospital and the rest of the determinations, the values of the day following fasting.

Laboratory analysis at the end of the study will be conducted with the patient 12 hours of fasting, before stopping the study medication.

Analyses were performed in the hospital laboratory Crossing according to standard techniques.

Assessing platelet aggregation was performed by aggregometry evaluated by turbidimetric method (AggRAM, Helena Laboratories, Beaumont, Texas, USA).

In tracking the value of blood pressure and heart rate were recorded at each visit, as well as pill counts were also conducted to assess adherence.

All data will be collected in a form designed for the study and stored in a database. The data input to the system will be performed to minimize duplicate entry errors in the information.

Follow up Follow-up visits will be conducted through interviews with one of the researchers.

The monitoring scheme is as follows:

* 7 days: an additional 7 days.
* At 30 days: an additional 15 days.
* At 3 months: an additional 15 days.
* At 6 months: an additional 15 days (final visit). Each visit will be an interview, physical examination and ECG. Counting capsules or pills to assess adherence is performed and a new supply of medication will be provided for the period until the next visit.

At the final visit, prior consultation with the researcher, a blood with 12 hours of fasting to corresponding laboratory evaluations will be performed.

Study Medication Study medication will be prepared in the hospital pharmacy Crossing protocolized according to procedures .

Losses to follow up Patients who did not attend one or more follow-up visits will be excluded from study analysis of adhesion. In all cases, telephone contact will attempt to determine the occurrence of adverse events.

Ethical Considerations Participants will be invited to participate in the study and will be explained in detail the objectives. Be given a copy of the written informed consent for their participation and can decide evacuate their doubts about the protocol.

The study was conducted according to the Declaration of Helsinki, the guidelines of international harmonization and local laws. In addition, the protocol will be conducted in accordance with the guidelines for good clinical practice.

They brighten at all times to patients the voluntary nature of participation in the study during the informed consent process. At each visit will be asked verbally about his desire to continue in the study.

Statistical Analysis Qualitative variables are described using numbers and percentages. Continuous variables were described using means and standard deviations or medians and interquartile ranges, if you have normal or non-normal distribution, respectively. Normality is determined by evaluating the quantile-quantile graphics and the Shapiro-Wilk test.

Analyses were performed according to the intention-to-treat analysis of all patients according to the group to which they were assigned.

The primary endpoint analysis was performed by Pearson chi2 test. Further estimate the relative risk of adhesion in the experimental treatment group compared to the control group, with their corresponding confidence intervals using a 2 x 2 table.

The differences between groups in levels of cholesterol and blood pressure were made using Student's t test.

Subgroup analyzes according to age (greater or less than the median), sex, education, diabetes, previous myocardial infarction and angioplasty was performed.

All analyzes were performed two-tailed and a p value less than 0.05 was used to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Myocardial infarction within seven (7) days prior: anginal symptoms with ST-segment changes (elevation or depression) or inversion of T waves or left bundle branch block and acute elevation of cardiac enzymes.
* Signature of written informed consent

Exclusion Criteria:

* Severe ventricular dysfunction, (ejection fraction of the left ventricle less than 40%)
* Contraindication for beta-blockers, angiotensin-converting enzyme, aspirin and / or statins.
* History of allergies or adverse reactions to some of the study drug reactions. Chronic treatment with NSAIDs. Planned coronary-revascularization within six months after discharge.
* Renal failure with estimated creatinine clearance according to the Cockroft-Gault formula less than 30 ml / min.
* Liver or elevated transaminases before randomization more than three times the upper normal limit.
* Higher fasting triglycerides 500 mg / dl.
* Indication according to medical criteria other than a beta-blocker atenolol.
* Indication of oral anticoagulation.
* Failure to follow due to difficulties of geographical access.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Adherence | Six months
  The adherence will be measures by pill count. It will presented as the percentage of pill taken on total theoretical pill that should be taken during the study period.

SECONDARY OUTCOMES:
Blood pressure, heart rate and cholesterol levels | Six months
  Measurement of blood pressure, heart rate and plasma levels of cholesterol.

OTHER OUTCOMES:
Platelet aggregation | Six months
  Measurement of platelet aggregation inhibition by aspirin. This outcome will be measured in a random subset of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Tajer, MD, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

REFERENCES:
- [Derived] Mariani J, Rosende A, De Abreu M, Gonzalez Villa Monte G, D'Imperio H, Antonietti L, Lemonnier G, de Bonis A, Tajer C. Multicap to improve adherence after acute coronary syndromes: results of a randomized controlled clinical trial. Ther Adv Cardiovasc Dis. 2020 Jan-Dec;14:1753944720912071. doi: 10.1177/1753944720912071. PMID 32186246